CLINICAL TRIAL: NCT04591236
Title: The Effect of Simultaneous Application of Transcranial Direct Current Stimulation (tDCS) and Gait Training for Parkinson's Disease Patients on Gait Function Improvement
Brief Title: Application of Transcranial Direct Current Stimulation (tDCS) for Gait Function Improvement of Parkinson's Disease Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-09-093
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: transcranial direct current stimulation; gait training; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait training with brain stimulation (Experimental): Treadmill gait training and transcranial direct current stimulation (tDCS) on the leg motor areas
  Interventions: Device: Brain stimulation; Device: Treadmill gait training
- Gait training with sham brain stimulation (Active Comparator): Treadmill gait training and anodal sham transcranial direct current stimulation (tDCS) on the leg motor areas
  Interventions: Device: Treadmill gait training

INTERVENTIONS:
Device: Brain stimulation — tDCS brain stimulation on leg motor areas was applied to Parkinson patients.
  Arms: Gait training with brain stimulation
Device: Treadmill gait training — Treadmill gait training was applied to Parkinson patients.

SUMMARY:
The purpose of this study was to investigate the effect of simultaneous application of transcranial direct current stimulation (tDCS) and treadmill gait training for gait function recovery in Parkinson's disease patients with gait impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50 - 75 years
* Modified Hoehn and Yahr stages 1 to 4

Exclusion Criteria:

* Serious cardiac conditions (hospitalization for myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living)
* Difficult to understand experimental tasks because of extremely severe cognitive impairment (Korean-Mini-Mental State Examination, K-MMSE≤10)
* History of psychiatric disease
* Implanted objects that would contraindicate tDCS

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Change in 10 meter walk test from baseline in gait speed | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)]
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

SECONDARY OUTCOMES:
Change in Berg Balance Scale (BBS) from baseline in balance | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)]
  Mesure of blance function. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Score the LOWEST performance. Total Score = 56.
Change in Timed Up and Go test (TUG) from baseline in balance | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)]
  Meserue of dynamic blance function. 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls.
Changes in Brain activation of resting-state functional MRI | session 0 (initial visit); session 10 (at approximately 4 weeks)
  Meserue of Neuroplasticity
Changes in motor evoked potentia | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)]
  Measure the motor threshold and amplitude of motor evoked potential in first dorsal interosseous muscle and TA muscle.
Changes in Functional Reach Test (FRT) from baseline | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)]
  FRT is a single item test developed as a quick screen for balance problems. Measurement Interpretation: 10"/25 cm or greater Low risk of falls; 6"/15cm to 10"/25cm Risk of falling is 2x greater than normal; 6"/15cm or less Risk of falling is 4x greater than normal; Unwilling to reach Risk of falling is 8x greater than normal
Change in muscle manual test (MMT) and range of motion (ROM) from baseline | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)]
  Meserue of MMT and ROM of lower extremity.
Change in Unified Parkinson's Disease Rating Scale (UPDRS) from baseline | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)]
  Meserue of Parkinson disease motor level.
  1) nonmotor experiences of daily living (13 items), (2) motor experiences of daily living (13 items), (3) motor examination (18 items), and (4) motor complications (six items). Each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.
Change in Korean Mini-Mental State Examination (K-MMSE) from baseline | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)]
  Meserue of cognition level. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age.
Change in Geriatric Depression Scale (GDS) from baseline | session 0 (initial visit); session 10 (at approximately 4 weeks); after 4 weeks from intervention termination (follow-up)]
  Meserue of depression. The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Lee, Ph.D, Principal Investigator — yun1225.kim@samsung.com
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided